CLINICAL TRIAL: NCT01276860
Title: The Use of Psychomotor Vigilance Testing in the Assessment of Pediatric Obstructive Sleep Apnea
Acronym: PVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 112316
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Results first posted 2020-06-12 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Pediatric Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Pediatric Obstructive Sleep Apnea; OSA; PVT; Psychomotor Vigilance Testing; Psychomotor Vigilance Task
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Psychomotor Vigilance Testing (Other): The purpose of this study is to examine the use of psychomotor vigilance testing (PVT) as a tool in the diagnosis and prediction of pediatric obstructive sleep apnea. PVT simply involves responding to a light by pressing a button on a small handheld device. It is a simple measure of reaction time.
  Interventions: Device: Psychomotor Vigilance Testing

INTERVENTIONS:
Device: Psychomotor Vigilance Testing — The purpose of this study is to examine the use of psychomotor vigilance testing (PVT) as a tool in the diagnosis and prediction of pediatric obstructive sleep apnea. PVT simply involves responding to a light by pressing a button on a small handheld device. It is a simple measure of reaction time.

SUMMARY:
Obstructive sleep apnea results in decreased attentiveness and response times in patients. The objective of this study is to quantify these consequences in pediatric OSA patients using an already established tool for examining the results of sleep deprivation and fragmentation: psychomotor vigilance testing. PVT has been used in children, but has not been studied in pediatric OSA patients. This study aims to employ PVT along the normal course of diagnosis and treatment of pediatric OSA patients in our clinical practice at Arkansas Children's Hospital. The investigators hypothesize that pediatric OSA patients will exhibit decreased PVT scoring when compared to children without OSA, and that PVT can be used to diagnose and monitor treatment outcomes in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pediatric patients ages 6-18 years old
* with symptoms of OSA (snoring, pauses in sleep breathing, restless sleep, frequent arousals, excellive daytime sleepiness, morning headaches)
* with physical exam findings consistent with adenotonsillar hypertrophy
* those identified as good candidates for adenotonsillectomy
* who are to undergo a polysomnogram as part of their preoperative work-up

Exclusion Criteria:

* History of attention deficit disorder, developmental delay, or mental retardation
* Children taking any neurotropic medications (including antiepileptics, antidepressives, and stimulants)
* Children previously treated for OSA (surgically or medically)
* Children with significant comorbidities including other sleep-related disorders

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gresham T Richter, MD, Principal Investigator — UAMS, ACH
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: PVT subjects with sleep complaints.
- Control Group: PVT subjects without sleep complaints.
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 5 | 2
Completed | 5 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: PVT subjects with sleep complaints.Control subjects will be asked to participate in one session. Treatment subjects will be asked to participate in 3 sessions.
- Control Group: PVT subjects without sleep complaints.Control subjects will be asked to participate in one session. Treatment subjects will be asked to participate in 3 sessions.
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Customized [Count of Participants; unit: Participants]
  6-18 years | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Criteria of Obstructive Sleep Apnea in the PVT Assessment
Description: Subjects with obstructive sleep apnea will be asked to participate in 3 sessions. Your child will be asked to complete some noninvasive tests at each session. These tests consist of Psychomotor Vigilance Task testing. A Psychomotor Vigilance Task (PVT) will measure your level of alertness and attentiveness. The PVT involves pressing a button after hearing a specific tone or seeing a flashing light. This test takes approximately 10 minutes to complete. The PVT testing will be done at the first clinic visit, then before any treatments, and finally after treatments have taken place. Outcome Measure is full completion of the PVT testing.
Time Frame: 10-20 minutes each session, 3 sessions total
Population: The analysis of each participant is based on the timing between hearing a specific tone or seeing a flashing light and the pressing of the button to record the alertness and attentiveness. Finalized analysis is not completed as the study was ended early and data not analyzed to compare groups.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Group: PVT subjects with sleep complaints/Obstructive Sleep Apnea.
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 5 | 2
Participants | 5 | 2

2. Secondary Outcome: Number of Participants Who Achieved Criteria of No Sleep Complaints in the PVT Assessment
Description: Subjects in the control group without clinical signs and symptoms of sleep apnea will only undergo PVT for one session. Your child will be asked to complete some noninvasive tests at this session. These tests consist of Psychomotor Vigilance Task testing. A Psychomotor Vigilance Task (PVT) will measure your level of alertness and attentiveness. The PVT involves pressing a button after hearing a specific tone or seeing a flashing light. This test takes approximately 10 minutes to complete. Outcome Measure is full completion of the PVT testing.
Time Frame: 10-20 minute session, 1 session
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 5 | 2
Participants | 5 | 2

ADVERSE EVENTS:
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 0/5 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No